CLINICAL TRIAL: NCT06914726
Title: Randomized Trial to Improve Care of Patients With Hereditary Cancer Syndromes
Brief Title: Patient Centered Clinical Decision Support for Hereditary Cancer Syndromes
Acronym: PC-CDS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-400; 1R01CA283332-01A1 (NIH)
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Hereditary Breast/Ovarian Cancer (brca1, brca2); Lynch Syndrome; Genetic Variation; HBOC Syndrome; Hereditary Cancer Syndromes
Keywords: Clinical Decision Support; Shared Decision Making; Hereditary Cancer Syndromes; Genetics; Genetic variations; HBOC; hereditary breast/ovarian cancer; BRCA1; BRCA2; Lynch Syndrome; Genetic variants
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome; Colorectal Neoplasms, Hereditary Nonpolyposis; Neoplastic Syndromes, Hereditary; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): All patients and clinicians at UC clinics will continue to receive an existing EHR-linked clinical decision support for management of major uncontrolled cardiovascular risk factors and other selected chronic conditions. The existing CDS displayed at UC clinics does not include patient-specific information on recommended cancer prevention activities for those with HBOC or LS.
- Patient Centered Clinical Decision Support for Hereditary Genetic Cancer Syndromes (Other): All patients and clinicians at PC-CDS clinics will continue to receive an existing EHR-linked clinical decision support for management of major uncontrolled cardiovascular risk factors and other selected chronic conditions plus patient-specific information on recommended cancer prevention activities for those with HBOC or LS.
  Interventions: Other: Patient Centered Clinical Decision Support (PC-CDS)

INTERVENTIONS:
Other: Patient Centered Clinical Decision Support (PC-CDS) — The intervention provides patient specific recommendations on managing cancer risk due to hereditary cancer gene variants that is integrated into an existing point of care clinical decision support system that algorithmically identifies study-eligible patients and deploys patient-specific CDS output at an index visit and all subsequent primary care encounters using the most up to date available clinical information.
  Other Names: Genetics Wizard
  Arms: Patient Centered Clinical Decision Support for Hereditary Genetic Cancer Syndromes

SUMMARY:
The goal of this clinical trial is to address care gaps for participants at high risk of breast and ovarian cancer (HBOC), or Lynch syndrome (LS) because of testing positive for specific genetic variants. A patient-centered clinical decision support (PC-CDS) tool will help identify participants with genetic variations and display recommendations for referrals and testing to the clinician and participant at a primary care visit. The main question the study aims to answer is:

- Does clinical decision support for participants with hereditary cancer syndromes improve the use of evidence-based cancer prevention care.

Participants being seen in the PC-CDS group are compared to participants being seen in usual care (UC) to see if they are up to date on guideline-based cancer prevention care and to see if participants in the PC-CDS group report more shared decision making and higher rates of self-management of their genetic cancer risks.

Participants will be asked to answer survey questions.

DETAILED DESCRIPTION:
Among the estimated one million Americans who have screened positive for specific genetic variants related to Hereditary Breast and Ovarian Cancer Syndrome (HBOC) or Lynch Syndrome (LS), less than half are up to date on evidence-based cancer prevention measures that may increase early detection of syndrome-related cancers or prevent these cancers altogether. Most patients newly diagnosed with hereditary cancer syndromes receive extensive initial care from genetic counselors or oncology teams but for many patients without a cancer diagnosis at the time of syndrome identification, access to regular follow-up care from oncologists and genetic counselors is limited. Pilot data show that the most frequent source of care for patients with HBOC or LS is the primary care setting, but many primary care clinicians (PCC) are unfamiliar with rapidly evolving cancer prevention guidelines for patients with HBOC or LS. Although PCCs are ideally positioned to make timely referrals to subspecialists for indicated cancer prevention care and procedures, access to evidence-based clinical decision support to optimize care for patients with these hereditary cancer syndromes does not exist.

PCCs provide care to over 80% of patients with HBOC or LS each year and are trained in shared decision making and coordination of care. However, the majority of PCCs are unaware of current recommendations for HBOC and LS and thus often fail to arrange appropriate referrals or procedures, including referrals to genetic counselors. The intervention targets these System and PCC-related barriers such as lack of awareness of the genetic condition, lack of knowledge of current evidence-based variant- specific care recommendations, and lack of timely referral for cancer prevention tests or procedures recommended for these high-risk patients. Both average-risk and high-risk patients are more likely to receive recommended cancer screening procedures when advised by their PCC.

The PC-CDS intervention also targets patient-related barriers to care, such as lack of awareness that certain tests or procedures are due, and lack of awareness of the benefits of certain interventions, tests, or procedures, and facilitates timely referral for access to subspecialists who can provide recommended services and procedures. Screening for CDC Tier 1 genetic conditions is rapidly increasing, but many of those who screen positive for HBOC or LS are not well-informed of evolving evidence-based care options. Current oncology teams are staffed primarily to deal with active management of cancer and have limited capacity to provide long-term care to large numbers of patients without diagnosed cancers. An estimated 33-50% of those diagnosed with these hereditary cancer syndromes do not complete a visit with a genetic counselor, with well-documented disparities in care for individuals with low income, low education, residence in inner city or rural areas, or membership in underserved racial/ethnic groups. Many patients with HBOC or LS are unaware of their risks, and the substantial health benefits obtainable by early detection and intervention; or lack the ability to coordinate their care across multiple subspecialists and care team members.

The PC- CDS provides each patient an updated list of variant-specific recommended care options and encourages and enables patients to have informed discussions of evidence-based care options with their PCCs or other trusted physicians. PCC referrals and suggestions will both directly and indirectly (through attitudes towards genetic conditions and intentions to access care) influence patient actions to adhere to evidence-based guidelines including (i) timely referrals to subspecialists (such as genetic counselors, oncologists, gastroenterologists, gynecologists, urologists, dermatologists, or surgeons) and (ii) engagement in recommended cancer prevention protocols and screening procedures.

This project provides evidence-based cancer prevention care recommendations to patients with HBOC or LS and their PCCs at primary care encounters when a given patient is not up to date on NCCN-recommended cancer prevention referrals and procedures. This specific application of health informatics technology to care of patients with these and other genetic variants is novel, in part because it relies on very recent advances in health informatics, increased rates of genetic screening within healthcare systems, and an accelerating (and rapidly evolving) knowledge base that supports an evidence-based set of variant-specific care recommendations. The intervention takes advantage of these recent developments and is designed to rapidly translate new genetic knowledge into evidence-based patient-specific clinical care. The variant-specific PC-CDS does not yet exist in primary care settings, and this project will provide a much-needed assessment of the impact of a PC-CDS intervention on cancer prevention care, shared decision making, and self-efficacy in managing hereditary cancer risks, as well as PCC knowledge of HBOC and LS cancer prevention care.

The web-based nature of the PC-CDS system, its prior success in improving primary care for a wide range of other chronic conditions, and its high use rates in primary care settings suggest that this approach to care improvement may be an effective strategy to increase appropriate referrals and evidence-based preventive care of adults with these hereditary cancer syndromes.

ELIGIBILITY:
Inclusion Criteria: The patient must meet all the following inclusion criteria on date of the Index Visit:

1. Aged 18 years or more at index clinical encounter,
2. Existing genetic testing or problem list evidence of HBOC or LS,
3. Index clinical encounter is with a PCC (family practice, general internal medicine, nurse practitioner, or physician assistant) at a randomized primary care clinic during the accrual period,
4. At the time of the index clinical encounter have EITHER (i) Evidence of having HBOC and not up-to- date on selected variant-specific cancer prevention care OR (ii) Evidence of having LS and not up-to-date on selected variant gene-specific cancer prevention care

Exclusion Criteria:

1. Diagnosis of dementia, OR
2. Currently receiving active treatment for cancer, OR
3. In long-term care, palliative care, or hospice care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2488 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Resolved care gaps | 18 months after index date
  Proportion of patients with a care gap for a specific genetic variant (HBOC: BRCA1, BRCA2; LS: MLH1, MSH2, MSH6, PMS2, or EPCAM) that is resolved within 18 months of index date.
Shared decision making | 12 months after index date
  Patient reports of shared decision making about their genetic risk using the Shared Decision-Making Questionnaire (SDM-Q-9) with total scores ranging from 0-45.
Self-eﬃcacy | 12 months after index date
  Patient reports of self-efficacy in managing cancer-related genetic risk using a modiﬁed version of the 12-item Communication and Attitudinal Self-Eﬃcacy scale for cancer (CASE-cancer) with scores ranging from 12-48.

SECONDARY OUTCOMES:
Resolved care gaps | 12 months after index date
  Proportion of patients with a care gap for a specific genetic variant (HBOC: BRCA1, BRCA2; LS: MLH1, MSH2, MSH6, PMS2, or EPCAM) that is resolved within 12 months of index date.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. O'Connor, MD, MPH, MA, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Medical Group, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Results of the study will be presented at local, regional, and national meetings and with HPMG leaders and leaders of other health care systems in the Twin Cities area. Results will also be published in peer-reviewed journals.
  The PC-CDS tool is Web-based, with potential for wide dissemination beyond HPMG. If permitted under then-current law, at the conclusion of the funding period, we plan to provide a de-identified data set to NCI for retention in a qualified data repository with appropriate mechanisms in place to guide the use of these data by other qualified researchers in the future.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Newton K, Green K, Lalloo F, Evans DG, Hill J. Colonoscopy screening compliance and outcomes in patients with Lynch syndrome. Colorectal Dis. 2015 Jan;17(1):38-46. doi: 10.1111/codi.12778. PMID 25213040
- [Background] Halbert CH, Lynch H, Lynch J, Main D, Kucharski S, Rustgi AK, Lerman C. Colon cancer screening practices following genetic testing for hereditary nonpolyposis colon cancer (HNPCC) mutations. Arch Intern Med. 2004 Sep 27;164(17):1881-7. doi: 10.1001/archinte.164.17.1881. PMID 15451763
- [Background] Daly MB, Pilarski R, Yurgelun MB, Berry MP, Buys SS, Dickson P, Domchek SM, Elkhanany A, Friedman S, Garber JE, Goggins M, Hutton ML, Khan S, Klein C, Kohlmann W, Kurian AW, Laronga C, Litton JK, Mak JS, Menendez CS, Merajver SD, Norquist BS, Offit K, Pal T, Pederson HJ, Reiser G, Shannon KM, Visvanathan K, Weitzel JN, Wick MJ, Wisinski KB, Dwyer MA, Darlow SD. NCCN Guidelines Insights: Genetic/Familial High-Risk Assessment: Breast, Ovarian, and Pancreatic, Version 1.2020. J Natl Compr Canc Netw. 2020 Apr;18(4):380-391. doi: 10.6004/jnccn.2020.0017. PMID 32259785
- [Background] Gabai-Kapara E, Lahad A, Kaufman B, Friedman E, Segev S, Renbaum P, Beeri R, Gal M, Grinshpun-Cohen J, Djemal K, Mandell JB, Lee MK, Beller U, Catane R, King MC, Levy-Lahad E. Population-based screening for breast and ovarian cancer risk due to BRCA1 and BRCA2. Proc Natl Acad Sci U S A. 2014 Sep 30;111(39):14205-10. doi: 10.1073/pnas.1415979111. Epub 2014 Sep 5. PMID 25192939
- [Background] Manickam K, Buchanan AH, Schwartz MLB, Hallquist MLG, Williams JL, Rahm AK, Rocha H, Savatt JM, Evans AE, Butry LM, Lazzeri AL, Lindbuchler DM, Flansburg CN, Leeming R, Vogel VG, Lebo MS, Mason-Suares HM, Hoskinson DC, Abul-Husn NS, Dewey FE, Overton JD, Reid JG, Baras A, Willard HF, McCormick CZ, Krishnamurthy SB, Hartzel DN, Kost KA, Lavage DR, Sturm AC, Frisbie LR, Person TN, Metpally RP, Giovanni MA, Lowry LE, Leader JB, Ritchie MD, Carey DJ, Justice AE, Kirchner HL, Faucett WA, Williams MS, Ledbetter DH, Murray MF. Exome Sequencing-Based Screening for BRCA1/2 Expected Pathogenic Variants Among Adult Biobank Participants. JAMA Netw Open. 2018 Sep 7;1(5):e182140. doi: 10.1001/jamanetworkopen.2018.2140. PMID 30646163
- [Background] Schneider KI, Schmidtke J. Patient compliance based on genetic medicine: a literature review. J Community Genet. 2014 Jan;5(1):31-48. doi: 10.1007/s12687-013-0160-2. Epub 2013 Aug 10. PMID 23934761
- See also: National Cancer Institute (n.d.), Evidence-Based Cancer Control Programs (EBCCP). Public Health Genomics Evidence-Based Programs Listing. — https://ebccp.cancercontrol.cancer.gov/topicPrograms.do?topicld=1196947&choice=default
- See also: National Cancer Institute. Cancer Stat Facts: Colorectal Cancer. Surveillance, Epidemiology and End Results Program — https://seer.cancer.gov/statfacts/html/colorect.html
- See also: Cancerwise — https://www.mdanderson.org/cancerwise.html